CLINICAL TRIAL: NCT04863612
Title: The Efficiency of SBRT in Preventing Recurrent Spinal Cord Compression in Patients Undergoing Surgery and Radiotherapy for Epidural Spinal Metastasis From Solid Tumor
Brief Title: SBRT in the Management of Solid Spinal Metastases
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: Extradural Tumors
Record Dates: First submitted 2021-02-19; First posted 2021-04-28 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-11

CONDITIONS: Extradural Tumor; Spinal Metastases
MeSH Terms: conditions — Epidural Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Documenting efficiency of SBRT in the management of epidural spinal metastases from solid tumors

DETAILED DESCRIPTION:
The department of radiotherapy in UZLeuven recently included Stereotactic Body Radiotherapy (SBRT) in the standard of care for the management of patients with spinal metastases. The aim of this study is to prospectively document neurological outcome, performance and quality of life following surgery + SBRT for spinal metastases with imminent / actual spinal cord compression, and compare outcomes with the historical cohort of the UZLeuven patients included in the Global Spine Tumor Study Group database between 2011 and 2019 in whom prospective neurological, performance and quality of life outcomes were collected following surgery + conventional radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Radiological diagnosis of spinal metastasis from solid tumor with epidural imminent or actual spinal cord compression, with or without neurological deficits. Patients will be scheduled for surgery + SBRT. If contra-indications preclude surgery and only SBRT is performed, patients will still be included.
* Written informed consent to participate in the study must be obtained from the subject or proxy /legal representative
* Males and females > 18 years

Exclusion Criteria:

* Any concomitant condition or disease which, in the opinion of the investigator, would affect the reliability of the collected data.
* Patients that had previous radiotherapy on the index spinal level without the possibility for additional SBRT at that particular level.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: males and females older then 18 years with radiological diagnosis of spinal metastais from solid tumor with epidural imminent or actual spinal cord compression with or without neurological deficits planned for surgery and SBRT.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2031-03-01 (Estimated); Study Completion 2036-03-01 (Estimated)

PRIMARY OUTCOMES:
neurological outcome Frankel scores | assessed up to 2 weeks prior to surgery
  Frankel scores (scale form A to E where A= complete loss of motor and sensory function, B= complete motor paralysis but some sensory function, C= some motor function but not usable, D= weakened but usable motor function, E= neurologically intact)
neurological outcome Frankel scores | assessed up to 2 weeks after surgery
  Frankel scores (scale form A to E where A= complete loss of motor and sensory function, B= complete motor paralysis but some sensory function, C= some motor function but not usable, D= weakened but usable motor function, E= neurologically intact)
neurological outcome Frankel scores | every 3 months, from date of surgery until date of decease or up to 1 year, whichever came first
  Frankel scores (scale form A to E where A= complete loss of motor and sensory function, B= complete motor paralysis but some sensory function, C= some motor function but not usable, D= weakened but usable motor function, E= neurologically intact)
neurological outcome Frankel scores | every year, from 1 year after surgery until date of decease or up to 5 years, whichever came first
  Frankel scores (scale form A to E where A= complete loss of motor and sensory function, B= complete motor paralysis but some sensory function, C= some motor function but not usable, D= weakened but usable motor function, E= neurologically intact)
neurological outcome Karnofsky score | assessed up to 2 weeks prior to surgery
  Karnofsky score (score from 100 to 10 where 100= no limitations, no complaints, 90= no limitations, minor symptoms, 80= no limitations, some symptoms, 70= care for himself, 60= requires occasional assistance, 50= considerable assistance/frequent care, 40= disabled, 30= severely disabled / hospitalisation, 20= very sick, hospitalisation, active support needed, 10= moribund)
neurological outcome Karnofsky score | assessed up to 2 weeks after surgery
  Karnofsky score (score from 100 to 10 where 100= no limitations, no complaints, 90= no limitations, minor symptoms, 80= no limitations, some symptoms, 70= care for himself, 60= requires occasional assistance, 50= considerable assistance/frequent care, 40= disabled, 30= severely disabled / hospitalisation, 20= very sick, hospitalisation, active support needed, 10= moribund)
neurological outcome Karnofsky score | every 3 months, from date of surgery until date of decease or up to 1 year, whichever came first
  Karnofsky score (score from 100 to 10 where 100= no limitations, no complaints, 90= no limitations, minor symptoms, 80= no limitations, some symptoms, 70= care for himself, 60= requires occasional assistance, 50= considerable assistance/frequent care, 40= disabled, 30= severely disabled / hospitalisation, 20= very sick, hospitalisation, active support needed, 10= moribund)
neurological outcome Karnofsky score | every year, from 1 year after surgery until date of decease or up to 5 years, whichever came first
  Karnofsky score (score from 100 to 10 where 100= no limitations, no complaints, 90= no limitations, minor symptoms, 80= no limitations, some symptoms, 70= care for himself, 60= requires occasional assistance, 50= considerable assistance/frequent care, 40= disabled, 30= severely disabled / hospitalisation, 20= very sick, hospitalisation, active support needed, 10= moribund)
neurological outcome urinary sphincter control | assessed up to 2 weeks prior to surgery
  based on patient reporting (normal, impaired, incontinent)
neurological outcome urinary sphincter control | assessed up to 2 weeks after surgery
  based on patient reporting (normal, impaired, incontinent)
neurological outcome urinary sphincter control | every 3 months, from date of surgery until date of decease or up to 1 year, whichever came first
  based on patient reporting (normal, impaired, incontinent)
neurological outcome urinary sphincter control | every year, from 1 year after surgery until date of decease or up to 5 years, whichever came first
  based on patient reporting (normal, impaired, incontinent)
performance and quality of life (EQ5D_3L) questionnaire | assessed up to 2 weeks prior to surgery
  data concerning mobility, self-care, usual activities, pain and discomfort, anxiety and depression will be collected
performance and quality of life (EQ5D_3L) questionnaire | assessed up to 2 weeks after surgery
  data concerning mobility, self-care, usual activities, pain and discomfort, anxiety and depression will be collected
performance and quality of life (EQ5D_3L) questionnaire | every 3 months, from date of surgery until date of decease or up to 1 year, whichever came first
  data concerning mobility, self-care, usual activities, pain and discomfort, anxiety and depression will be collected
performance and quality of life (EQ5D_3L) questionnaire | every year, from 1 year after surgery until date of decease or up to 5 years, whichever came first
  data concerning mobility, self-care, usual activities, pain and discomfort, anxiety and depression will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Bart Depreitere, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- University hospital Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No